CLINICAL TRIAL: NCT03726385
Title: Investigation of the Effectiveness of Visual Feedback Training on Upper Extremity Functions
Brief Title: Investigation of the Effectiveness of Visual Feedback Training on Upper Extremity Functions in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Dilara Merve Sarı (Other)
Responsible Party: Sponsor-Investigator, Dilara Merve Sarı, Director of Physiotherapy Department, Dilbade Education and Rehabilitation Center
Organization: Dilbade Education and Rehabilitation Center (Other)
Other Study IDs: DilbadeEdRehabCtr
Record Dates: First submitted 2018-10-27; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; upper extremity rehabilitation; neurodevelopmental therapy; physiotherapy and rehabilitation; visual feedback device
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Group I: The control group. Participants in this group received only NDT based upper extremity rehabilitation. Number of the participants were 19.
- Group II: Group II: The study group. Participants in this group received NDT based upper extremity rehabilitation + Cogniboard® Light Trainer training. Number of the participants were 19.

SUMMARY:
The purpose of the study was to investigate the effectiveness of Cogniboard® Light Trainer, an education device with visual feedback that is added to the Neurodevelopmental Therapy Method (NDT) based upper extremity rehabilitation in children with cerebral palsy, on upper extremity functions such as joint range of motion (ROM), muscle tone, grip strength, pinch strength and functional abilities.

DETAILED DESCRIPTION:
Children with the diagnosis of Cerebral Palsy, aged between 4 and 18 years were included in the study, who were volunteered to participate. The participants were randomly assigned into two groups; A total of 16 sessions of rehabilitation program were applied for 2 days a week for 8 weeks. The treatment programs applied are; Group I: NDT based upper extremity rehabilitation, Group II: NDT based upper extremity rehabilitation + Cogniboard® Light Trainer training. In the cases, pre- and post-treatment spasticity was defined with 'Modified Ashworth Scale'; upper extremity joint range of motion (ROM) with 'goniometer'; grip and pinch strength with 'dynamometer'; hand skills with 'Minnesota Hand Skill Test'; functional abilities with 'Childhood Health Assessment Questionnaire (CHAQ) and functional level with 'Gross Motor Function Classification System (GMFCS)'.

ELIGIBILITY:
Inclusion Criteria:

* Having the diagnosis of Cerebral Palsy (CP),
* Aged between 4-18,
* Having 1+ upper extremity spasticity at max according to the Modified Ashworth Scale (MAS),
* To be able to cooperate with exercises

Exclusion Criteria:

* Having mental retardation report,
* Having congenital deformities,
* Epilepsy history,
* Having cardiac, orthopedic, visual and hearing problems,
* Application of Botulinum Toxin (BOTOX) to the upper extremity in past six month.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants of the study were selected among the children who applied to Dilbade Education and Rehabilitation Center for rehabilitation.
  Simple random sampling method was applied to group selection.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM) | Eight weeks
  Upper extremity ROM measured with universal goniometer.
Spasticity | Eight weeks
  Spasticity defined with Modified Ashworth Scale (MAS). The MAS measures resistance during passive soft-tissue stretching. Scoring: 0= normal tone. 1= slight increase in muscle tone, minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion or extension. 1+= slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder of the ROM. 2= more marked increase in muscle tone through most of the ROM, but affected part(s) easily moved. 3= considerable increase in muscle tone, passive movement difficult. 4= affected part(s) rigid in flexion or extension.
Grip and pinch strength | Eight weeks
  Grip and pinch strength measured with dynamometer.
Hand Skills | Eight weeks
  Hand skills was assessed with Minnesota Dexterity Test (MMDT). MMDT is a standardized test for the evaluation of a subject's ability to move small objects various distances. The score on the test is the total seconds required to complete chosen number of test trials.
Functional Abilities | Eight weeks
  Functional abilities was assessed with Childhood Health Assessment Questionnaire (CHAQ). CHAQ is used to assess health status in children. It assesses functional ability in 8 domains of physical function (30 items) for children. Each item is scored on a four point scale ranging from 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), 3 (unable to do). The mean score of the eight domains finally makes up the disability index and ranges from 0 (no disability) to 3 (disabled).
Functional Level | Eight weeks
  Functional level was defined with Gross Motor Function Classification System (GMFCS). GMFCS looks at movements such as sitting, walking and use of mobility devices. It provides a clear description of a child's current gross motor function. Level I can climb stairs without the use of a railing. Level II can walk in most settings and climb stairs holding onto a railing. Level III needs usage of a hand held mobility device, may climb stairs holding onto a railing with assistance. Level IV requires physical assistance or powered mobility in most settings. Level V children are transported in a manuel wheelchair in all settings, they are limited in their ability to maintain antigravity head and trunk postures and control leg and arm movements.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Kuru Colak, Study Director — Marmara University Institute of Health Sciences
Locations (1):
- Dilbade Education and Rehabilitation Center, Istanbul, Eyup, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR) might be considered to be shared with clinicians studying in the same field one year after the publication of the study.

REFERENCES:
- [Background] Acar G, Altun GP, Yurdalan S, Polat MG. Efficacy of neurodevelopmental treatment combined with the Nintendo((R)) Wii in patients with cerebral palsy. J Phys Ther Sci. 2016 Mar;28(3):774-80. doi: 10.1589/jpts.28.774. Epub 2016 Mar 31. PMID 27134357
- [Background] Avery LM, Russell DJ, Raina PS, Walter SD, Rosenbaum PL. Rasch analysis of the Gross Motor Function Measure: validating the assumptions of the Rasch model to create an interval-level measure. Arch Phys Med Rehabil. 2003 May;84(5):697-705. doi: 10.1016/s0003-9993(02)04896-7. PMID 12736885
- [Background] Yam WK, Leung MS. Interrater reliability of Modified Ashworth Scale and Modified Tardieu Scale in children with spastic cerebral palsy. J Child Neurol. 2006 Dec;21(12):1031-5. doi: 10.1177/7010.2006.00222. PMID 17156693
- [Background] James S, Ziviani J, Ware RS, Boyd RN. Relationships between activities of daily living, upper limb function, and visual perception in children and adolescents with unilateral cerebral palsy. Dev Med Child Neurol. 2015 Sep;57(9):852-7. doi: 10.1111/dmcn.12715. Epub 2015 Feb 23. PMID 25703777
- [Background] Gilliaux M, Renders A, Dispa D, Holvoet D, Sapin J, Dehez B, Detrembleur C, Lejeune TM, Stoquart G. Upper limb robot-assisted therapy in cerebral palsy: a single-blind randomized controlled trial. Neurorehabil Neural Repair. 2015 Feb;29(2):183-92. doi: 10.1177/1545968314541172. Epub 2014 Jul 11. PMID 25015650
- [Background] Chiu HC, Ada L, Lee HM. Upper limb training using Wii Sports Resort for children with hemiplegic cerebral palsy: a randomized, single-blind trial. Clin Rehabil. 2014 Oct;28(10):1015-24. doi: 10.1177/0269215514533709. Epub 2014 May 21. PMID 24849793
- [Background] Hutzler Y, Lamela Rodriguez B, Mendoza Laiz N, Diez I, Barak S. The effects of an exercise training program on hand and wrist strength, and function, and activities of daily living, in adults with severe cerebral palsy. Res Dev Disabil. 2013 Dec;34(12):4343-54. doi: 10.1016/j.ridd.2013.09.015. Epub 2013 Oct 18. PMID 24145046
- [Background] Klimont L. Principles of Bobath neuro-developmental therapy in cerebral palsy. Ortop Traumatol Rehabil. 2001;3(4):527-30. PMID 17984909
- [Background] Klingels K, De Cock P, Molenaers G, Desloovere K, Huenaerts C, Jaspers E, Feys H. Upper limb motor and sensory impairments in children with hemiplegic cerebral palsy. Can they be measured reliably? Disabil Rehabil. 2010;32(5):409-16. doi: 10.3109/09638280903171469. PMID 20095955
- [Background] Koman LA, Williams RM, Evans PJ, Richardson R, Naughton MJ, Passmore L, Smith BP. Quantification of upper extremity function and range of motion in children with cerebral palsy. Dev Med Child Neurol. 2008 Dec;50(12):910-7. doi: 10.1111/j.1469-8749.2008.03098.x. Epub 2008 Sep 20. PMID 18811712
- [Background] MacIntosh A, Lam E, Vigneron V, Vignais N, Biddiss E. Biofeedback interventions for individuals with cerebral palsy: a systematic review. Disabil Rehabil. 2019 Oct;41(20):2369-2391. doi: 10.1080/09638288.2018.1468933. Epub 2018 May 12. PMID 29756481
- [Background] Narayanan UG. The role of gait analysis in the orthopaedic management of ambulatory cerebral palsy. Curr Opin Pediatr. 2007 Feb;19(1):38-43. doi: 10.1097/MOP.0b013e3280118a6d. PMID 17224660
- [Background] Ozdogan H, Ruperto N, Kasapcopur O, Bakkaloglu A, Arisoy N, Ozen S, Ugurlu U, Unsal E, Melikoglu M; Paediatric Rheumatology International Trials Organisation. The Turkish version of the Childhood Health Assessment Questionnaire (CHAQ) and the Child Health Questionnaire (CHQ). Clin Exp Rheumatol. 2001 Jul-Aug;19(4 Suppl 23):S158-62. PMID 11510322
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Park EY, Kim WH. Effect of neurodevelopmental treatment-based physical therapy on the change of muscle strength, spasticity, and gross motor function in children with spastic cerebral palsy. J Phys Ther Sci. 2017 Jun;29(6):966-969. doi: 10.1589/jpts.29.966. Epub 2017 Jun 7. PMID 28626301
- [Background] Plautz EJ, Milliken GW, Nudo RJ. Effects of repetitive motor training on movement representations in adult squirrel monkeys: role of use versus learning. Neurobiol Learn Mem. 2000 Jul;74(1):27-55. doi: 10.1006/nlme.1999.3934. PMID 10873519
- [Background] Ravi DK, Kumar N, Singhi P. Effectiveness of virtual reality rehabilitation for children and adolescents with cerebral palsy: an updated evidence-based systematic review. Physiotherapy. 2017 Sep;103(3):245-258. doi: 10.1016/j.physio.2016.08.004. Epub 2016 Sep 27. PMID 28109566
- [Background] Rosenbaum PL, Palisano RJ, Bartlett DJ, Galuppi BE, Russell DJ. Development of the Gross Motor Function Classification System for cerebral palsy. Dev Med Child Neurol. 2008 Apr;50(4):249-53. doi: 10.1111/j.1469-8749.2008.02045.x. Epub 2008 Mar 1. PMID 18318732
- [Background] Ruperto N, Ravelli A, Pistorio A, Malattia C, Cavuto S, Gado-West L, Tortorelli A, Landgraf JM, Singh G, Martini A; Paediatric Rheumatology International Trials Organisation. Cross-cultural adaptation and psychometric evaluation of the Childhood Health Assessment Questionnaire (CHAQ) and the Child Health Questionnaire (CHQ) in 32 countries. Review of the general methodology. Clin Exp Rheumatol. 2001 Jul-Aug;19(4 Suppl 23):S1-9. PMID 11510308
- [Background] Saposnik G, Mamdani M, Bayley M, Thorpe KE, Hall J, Cohen LG, Teasell R; EVREST Steering Committee; EVREST Study Group for the Stroke Outcome Research Canada Working Group. Effectiveness of Virtual Reality Exercises in STroke Rehabilitation (EVREST): rationale, design, and protocol of a pilot randomized clinical trial assessing the Wii gaming system. Int J Stroke. 2010 Feb;5(1):47-51. doi: 10.1111/j.1747-4949.2009.00404.x. PMID 20088994
- [Background] Serdaroglu A, Cansu A, Ozkan S, Tezcan S. Prevalence of cerebral palsy in Turkish children between the ages of 2 and 16 years. Dev Med Child Neurol. 2006 Jun;48(6):413-6. doi: 10.1017/S0012162206000910. PMID 16700929
- [Background] Shechtman O, Gestewitz L, Kimble C. Reliability and validity of the DynEx dynamometer. J Hand Ther. 2005 Jul-Sep;18(3):339-47. doi: 10.1197/j.jht.2005.04.002. PMID 16059855
- [Background] Spittle AJ, Doyle LW, Boyd RN. A systematic review of the clinimetric properties of neuromotor assessments for preterm infants during the first year of life. Dev Med Child Neurol. 2008 Apr;50(4):254-66. doi: 10.1111/j.1469-8749.2008.02025.x. Epub 2008 Jan 7. PMID 18190538
- [Background] Tesio L, Simone A, Zebellin G, Rota V, Malfitano C, Perucca L. Bimanual dexterity assessment: validation of a revised form of the turning subtest from the Minnesota Dexterity Test. Int J Rehabil Res. 2016 Mar;39(1):57-62. doi: 10.1097/MRR.0000000000000145. PMID 26579699
- [Background] Tredgett MW, Davis TR. Rapid repeat testing of grip strength for detection of faked hand weakness. J Hand Surg Br. 2000 Aug;25(4):372-5. doi: 10.1054/jhsb.2000.0433. PMID 11058007
- [Background] Zoccolillo L, Morelli D, Cincotti F, Muzzioli L, Gobbetti T, Paolucci S, Iosa M. Video-game based therapy performed by children with cerebral palsy: a cross-over randomized controlled trial and a cross-sectional quantitative measure of physical activity. Eur J Phys Rehabil Med. 2015 Dec;51(6):669-76. Epub 2015 Feb 5. PMID 25653079

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03726385/Prot_SAP_ICF_000.pdf